CLINICAL TRIAL: NCT03506425
Title: A Pilot Trial of Triheptanoin for People With Amyotrophic Lateral Sclerosis (PALS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Richard Bedlack, M.D., Ph.D. (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Richard Bedlack, M.D., Ph.D., MD, PhD, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00092250
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: ALS
MeSH Terms: interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Standard care for 1 month, then standard care and Triheptanoin for 5 months.
  Interventions: Drug: Triheptanoin
- Group 2 (Experimental): Standard care and Triheptanoin for 6 months.
  Interventions: Drug: Triheptanoin
- Group 3 (No Intervention): Healthy controls for biomarkers

INTERVENTIONS:
Drug: Triheptanoin — Triheptanoin is a medium chain triglyceride (MCT) that can improve mitochondrial function and energy production and therefore has potential for slowing ALS progression. Indeed, triheptanoin slowed motor neuron loss and delayed the onset of weakness in a mutant SOD1 model of ALS. The Triheptanoin we will use is a colorless to light yellow oil. The target triheptanoin dose for this study is 1g/kg/d. This target dose was selected because it was safe and tolerable and altered brain MR spectroscopy in patients with Huntington's Disease.
  Arms: Group 1; Group 2

SUMMARY:
The causes of ALS are largely unknown. However, mitochondrial dysfunction, resulting in impaired energy production, oxidative stress and apoptosis, may play a key role in ALS progression. Triheptanoin can improve mitochondrial function and energy production and therefore has potential for slowing ALS progression. Indeed, triheptanoin slowed motor neuron loss and delayed the onset of weakness in a mutant SOD1 model of ALS. This pilot trial will determine if Triheptanoin is safe tolerable, alters biomarkers of brain energy metabolism and oxidative stress, and slows functional decline in people with ALS.

DETAILED DESCRIPTION:
This is an open label, prospective cohort study of 10 people with ALS (PALS) from the Duke ALS Clinic. The first 5 enrolled PALS (Group 1) will receive standard ALS care for the first month, then standard care plus Triheptanoin for the next 5 months. The next 5 enrolled PALS (Group 2) will receive standard ALS care plus Triheptanoin for 6 months (Figure 1). All Group 1 and Group 2 PALS who complete this 6-month study will have an option for Triheptanoin treatment extension for an additional 12 months. In addition to the PALS, there will also be 5 healthy controls enrolled (Group 3), people that do not have ALS or any other neurodegenerative disease). These participants will not receive any treatment; the only outcome measure they will complete is serum and urine biomarker testing at screening/baseline, month 1 and month 6.

The rationale for delaying triheptanoin treatment in one group is to look for differences in MR spectroscopy related to treatment at the 1 month time point. The target triheptanoin dose for this study is 1g/kg/d. This target dose was selected because it was safe and tolerable and altered brain MR spectroscopy in patients with Huntington's Disease. Participants will taper up to this dose as follows: start at 0.25g/kg/d for 1 week, then take 0.5g/kg/d for 1 week, then take 1g/kg/d and stay on this dose for the duration of the study. Triheptanoin will be administered orally with food or by gastrostomy tube over 3 divided doses (breakfast, lunch, and dinner). If at any point after week 1 a participant does not appear to be tolerating their current dose, it will be reduced by 0.25g/kg/d. If they cannot tolerate the starting dose of 0.25g/kg/d, the treatment will be discontinued. A dietician will make contact with all participants every month, either in person or by telephone, to try and maximize compliance.

The primary outcome measure is the ALSFRS-R score obtained monthly for all treated participants (in person at screening/baseline, month 1, month 3 and month 6; via telephone at months 2, 4 and 5). We will also obtain this measure by phone at months 6 and 12 of the extension. For all enrolled PALS in Groups 1 and 2, we will compare the slope of ALSFRS-R progression before enrollment to the slop of ALSFRS-R progression during the trial. ALSFRS-R is a quickly administered (five minute) ordinal rating scale (ratings 0-4) used to determine patients' assessments of their capability and independence in 13 functional activities. All 13 activities are relevant in ALS. Initial validity was established in ALS patients by documenting that their change in ALSFRS-R scores, which correlated with change in strength over time, was closely associated with quality of life measures, and predicted survival. The test-retest reliability is greater than 0.88 for all 13 itemsactivities. The ALSFRS-R declines linearly with time over a wide range during the course of ALS. The minimum clinically significant change in this scale is said to be 20%. The measure can be reliably conducted over the phone.

Secondary outcome measures include:

MR Spectroscopy NAA/Cr ratio in motor cortex will be measured at screening/baseline and 1 month time points. This measure declines over time in patients with ALS. This measure can respond to treatment; it was shown to improve over 3 weeks in patients with ALS on riluzole compared to a group that was not on this treatment. We will compare the MR spectroscopy changes over 1 month in Group 1 to the MR spectroscopy changes over 1 month in Group 2.

A Serum and Urine Biomarker Panel will be obtained at screening/baseline, 1 month and 6-month time points and analyzed using liquid chromatography/tandem mass spectrometry. Laboratory, pathologic, and epidemiologic evidence clearly supports the hypothesis that oxidative stress is central in the ALS pathogenic process, particularly in genetically susceptive individuals. Oxidative stress biomarkers in cerebrospinal fluid, plasma, and urine are elevated, suggesting that abnormal oxidative stress is generated outside of the central nervous system. Magnitude of lipid peroxidation, measured as non-enzymatic oxidation products of arachidonic acid, F2-isoprostanes, appears the most obvious oxidative stress marker. We will measure urine F2-isoprostane metabolites (class III: iPF2α-III, and 2,3-dinor iPF-2alpha-III, class VI: iPF-2alpha-VI, and 8,12-iso-iPF-2alpha-VI), urine creatinine, and serum and urine glutamate, a-keto-glutarate, NADH, coenzyme A levels in all treated participants and healthy controls at screening/baseline, month 1 and month 6 time points. We will compare the biomarker changes at different times points across between Groups 1, 2 and 3.

For safety monitoring:, concomitant medications, vital signs, weight, physical exam and safety labs (CBC, CMP, Lipid Profile, GGT, LFT and pregnancy testing for sexually active females with child bearing potential) will be measured at screening/baseline, 1 month, 3 month, and 6-month time points. Adverse events will be monitored continuously throughout the study, as described in Section 5.1.

The primary statistical analysis is the slope of the revised ALS functional rating scale (ALSFRS-R) during treatment compared to pre-treatment. Pre-treatment slope for each participant will be estimated as follows: (48-enrollment ALSFRS-R)/months since symptom onset. This frequently used "pre-slope" method is simple and inexpensive, and can predict disease progression as well as more complicated and expensive tools, at least for periods of less than 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Lab supported probable or more definite ALS by El Escorial Criteria
2. Age greater than or equal to 18 years
3. Willing and able to provide informed consent
4. On riluzole at a stable dose for at least 30d or not taking this
5. On Radicava at a stable dose for at least 30d or not taking this
6. Life expectancy at least 6 months
7. Currently managed on a reasonably stable diet, avoidance of fasting, carnitine or medium chain triglyceride (MCT) oils
8. Must stop any other experimental ALS treatment for at least 30 days prior to screening
9. If sexually active, must agree to use contraceptive or abstinence for duration of treatment with triheptanoin
10. Females of child bearing age must have negative pregnancy test at screening

Exclusion Criteria:

1. Unwilling or unable to provide informed consent
2. Previous intolerance or adverse reaction to triheptanoin or MCT
3. Conditions that will prohibit MRI scanning (metal in eye, some surgical implants, claustrophobia, inability to lie supine)
4. Have any other co-morbid conditions that in the opinion of the study investigator, places the participant at increased risk of complications, interferes with study participation or compliance, or confounds study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bedlack, MD PhD, Principal Investigator — Duke ALS Clinic
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data from this small pilot trial

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 5 | 5 | 5
Completed | 3 | 2 | 4
Not Completed | 2 | 3 | 1
Not completed — Adverse Event | 1 | 3 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.3) | 59.0 (14.4) | 55.6 (14.4) | 57.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 5 | 6
  Male | 5 | 4 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 4 | 4 | 5 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: ALS Functional Rating Scale-revised Version (ALSFRS-R) Slope
Description: Amyotrophic lateral sclerosis functional rating scale-revised version (ALSFRS-R) is used to determine patients' assessments of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS and each is scored between 0 (no function at all) and 4 (normal function). Thus the overall score for this measure can range from 0 to 48, with higher scores indicating more normal function. The test-retest reliability is greater than 0.88 for all 12 items/activities. The ALSFRS-R declines linearly with time over a wide range during the course of ALS and the minimum clinically significant change in this scale is said to be 20%. The primary analysis in this study is the slope of the ALSFRS-R during treatment compared to pre-treatment. Pre-treatment slope for each participant will be estimated as follows: (48-enrollment ALSFRS-R)/months since symptom onset. This frequently used "pre-slope" method is simple and inexpensive, and can predict disease progression.
Time Frame: baseline, 6 months
Population: For the primary outcome measure, patients in Arm 1 and Arm 2 were combined (since patients in both these groups received at least 5 months of Triheptanoin). The primary outcome comparison is not between these arms, but between all these Triheptanoin-treated patients' ALSFRS-R progression during the study compared to progression before the study.
Measure: Mean (Standard Deviation); unit: points per month
Groups:
- All Completed Subjects - Groups 1 and 2: Group 1: Standard care for 1 month, then standard care and Triheptanoin for 5 months.
  Group 2: Standard care and Triheptanoin for 6 months.
  Triheptanoin: Triheptanoin is a medium chain triglyceride (MCT) that can improve mitochondrial function and energy production and therefore has potential for slowing ALS progression. Indeed, triheptanoin slowed motor neuron loss and delayed the onset of weakness in a mutant SOD1 model of ALS. The Triheptanoin we will use is a colorless to light yellow oil. The target triheptanoin dose for this study is 1g/kg/d. This target dose was selected because it was safe and tolerable and altered brain MR spectroscopy in patients with Huntington's Disease.
Arm/Group | All Completed Subjects - Groups 1 and 2
Number analyzed (Participants) | 5
points per month
  ALSFRS-R During Treatment | -0.39 (0.44)
  ALSFRS-R Before Treatment | -0.57 (0.43)
Statistical Analysis 1: Comparison: All Completed Subjects - Groups 1 and 2; Test type: Other; p = 0.32, t-test, 2 sided

2. Secondary Outcome: Change in NAA/Cr Ratio From Motor Cortex as Measured by Magnetic Resonance Spectroscopy
Description: Effects of time, Triheptanoin on NAA/Cr (N-acetylaspartate/creatine) ratio from motor cortex
Time Frame: baseline, 6 months
Population: One subject in Group 2 did not complete the second MRS measure. Group 3 did not receive treatment; therefore, no data was collected on Group 3 for this outcome measure.
Measure: Mean (Standard Deviation); unit: NAA/Cr
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 4
NAA/Cr | 0.4188 (0.1923) | 0.0875 (0.3013)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Other; p = 0.08, ANOVA

3. Secondary Outcome: Change in Urine Isoprostane Levels, an Oxidative Stress Marker
Description: Effects of ALS and/or Triheptanoin on urine isoprostane levels (a marker of oxidative stress) at month 1
Time Frame: baseline, 1 month
Population: One subject in Group 2 did not complete the month 1 visit.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 5 | 4 | 5
ng/mg | 0.33 (0.38) | 0.32 (0.10) | 0.26 (0.12)
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Other; p = 0.83, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=5) | Group 2 (N=5) | Group 3 (N=5)
Death (Nervous system disorders) | 1 | 0 | 0
Hypercarbic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=5) | Group 2 (N=5) | Group 3 (N=5)
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Anorexia (Gastrointestinal disorders) | 1 | 1 | 0
Weight gain (Gastrointestinal disorders) | 1 | 1 | 0
Weight loss (Gastrointestinal disorders) | 1 | 0 | 0
Stomach cramps (Gastrointestinal disorders) | 0 | 2 | 0
Increased AST and ALT (Gastrointestinal disorders) | 0 | 1 | 0
Leg pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Hoarseness (Nervous system disorders) | 1 | 1 | 0
Fatigue (Nervous system disorders) | 0 | 2 | 0
Vertigo (Nervous system disorders) | 0 | 1 | 0
Increased weakness (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT03506425/Prot_SAP_000.pdf